CLINICAL TRIAL: NCT02526225
Title: A Randomized,Double Blind,Placebo Parallel Controlled,Multicenter Clinical Sthdy of Ginkgo Diterpene Lactone Meglumine Injection for Acute Ischemic Stroke Efficacy Safety.
Brief Title: A Safety and Effective Study of Ginkgolides Diterpene Lactone Meglumine Injection in the Treatment of Ischemic Stroke.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Bionovo Medicine Development Co., Ltd. (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Executive Vice-President, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1412-Z-YXET-ZS-RE
Record Dates: First submitted 2015-08-05; First posted 2015-08-18 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Ischemic Stroke
Keywords: acute ischemic stroke; safety and effectiveness; Ginkgo diterpene lactone meglumine injection
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ginkgo diterpene lactone meglumine injection (Active Comparator): ginkgo diterpene lactone meglumine injection
  Interventions: Drug: Ginkgo diterpene lactone meglumine injection
- Ginkgo diterpene lactone meglumine injection simulation (Placebo Comparator): Ginkgo diterpene lactone meglumine injection simulation
  Interventions: Drug: Ginkgo diterpene lactone meglumine injection simulation

INTERVENTIONS:
Drug: Ginkgo diterpene lactone meglumine injection — 5 ml/times, 1 time/day.Before use, the drug slowly added to the 0.9% sodium chloride injection diluted in 250 ml, slow intravenous drip.
  Arms: ginkgo diterpene lactone meglumine injection
Drug: Ginkgo diterpene lactone meglumine injection simulation — 5 ml/times, 1 time/day.Before use, the drug slowly added to the 0.9% sodium chloride injection diluted in 250 ml, slow intravenous drip.
  Arms: Ginkgo diterpene lactone meglumine injection simulation

SUMMARY:
The aim of this study is to evaluate the safety and effectivity of Ginkgo diterpene lactone meglumine injection tn the treatment of acute ischemic stroke

DETAILED DESCRIPTION:
After randomized to 90 + 7 days mRS 0-1 points is the Primary Outcome Measure,evaluate the safety and effectivity of Ginkgo diterpene lactone meglumine injection tn the treatment of acute ischemic stroke

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years of age, and gender not limited。
2. Within 48 hours of stroke onset of ischemic stroke (diagnosis standard by the Chinese medical association of the fourth national conference on cerebrovascular disease);
3. The first onset, or always not obvious legacy of stroke sequela (mRS acuities were before the onset of 1);
4. The degree of nerve function defect score (NIHSS) score 4 to 24 points, body movement component (NIHSS score paragraphs 5 and 6) total score 2 points or higher;
5. Understand and voluntarily signed informed consent.

Exclusion Criteria:

1. Head imaging studies have confirmed that, encephalitis, brain tumor, brain abscess and cause similar symptoms of disease, or confirm with hemorrhagic cerebral infarction, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, etc.
2. The serious disturbance of consciousness (Ia NIHSS score 2 points or higher);
3. With hemorrhagic disease or have a bleeding tendency, or have a lower limb venous thrombosis;
4. Serious abnormal liver and kidney function, liver function laboratory indexes of ALT > 3 ULN, renal laboratory ULN Cr > 1.5);
5. A history of mental illness or dementia patients;
6. Severe organ or other systemic disease, accompanied by any organ or system of malignant tumor, or ongoing anti-tumor treatment, the estimated lifetime < 3 months;
7. Significant drug or alcohol abuse;
8. Allergic constitution, as well as to two or more drugs or food allergies;This medicine ingredients allergy or known;
9. Have pregnancy (check blood HCG positive screening tests, namely HCG > 5 miu/mL), during the test preparation is pregnancy or lactation in women;
10. In the past three months in other clinical trials;
11. Researchers do not determine poor adherence, or any other suitable for patients to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3452 (Actual)
Dates: Start 2016-02-01; Primary Completion 2018-05-01 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Modified Rankin Scale (mRS) less than or equal to 1 . | 90 days

SECONDARY OUTCOMES:
Proportion of patients with National Institutes of Health Stroke Score (NIHSS) rising 4 or more points, three points, two points, one of the subjects changes from baseline to randomized 7 days. | Baseline, 7days
Proportion of patients with National Institutes of Health Stroke Score (NIHSS) reducing 4 points or more changes from baseline to randomized 7 days,14 days. | Baseline,7 days,14 days,
Proportion of patients with Modified Rankin Scale (mRS) reaching 0-2 . | 90 days
The Montreal Cognitive Assessment (MoCA) scale changes from baseline to randomized 14 days,90 days. | Baseline,14 days,90 days
The EuroQol-5 Dimensions (EQ-5D) scale changes from baseline to randomized 14 days,90 days. | Baseline,14 days,90 days
The all-cause mortality | 90 days
Ischemic stroke recurrence rate | 90 days
Composite incidence of vascular events | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: yongjun wang, M.D., Principal Investigator — Beijing Tiantan Hospital,Capital Medical University,Bgeijing,China
Locations (1):
- Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Tian X, Xu Q, Xia X, Zhang Y, Zhao X, Wang A. Effect of ginkgo diterpene lactone meglumine on the quality of life in patients with acute ischemic stroke. Health Qual Life Outcomes. 2024 Nov 15;22(1):99. doi: 10.1186/s12955-024-02315-1. PMID 39548582
- [Derived] Zhang Q, Wang A, Xu Q, Xia X, Tian X, Zhang Y, Li X, Yang X, Wang X, Peng J, Li Y, Liu L, Jin S, Meng X, Zhao X; GDLM group. Efficacy and Safety of Ginkgo Diterpene Lactone Meglumine in Acute Ischemic Stroke: A Randomized Clinical Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2328828. doi: 10.1001/jamanetworkopen.2023.28828. PMID 37578791